CLINICAL TRIAL: NCT06724315
Title: Prospective and Multicentric Cohort Study of Severe and Very Severe Chronic Obstructive Pulmonary Disease (COPD) in Brazil (SCOPe).
Acronym: SCOPe
Status: Recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: SCOPe
Record Dates: First submitted 2024-11-18; First posted 2024-12-09 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; Exacerbation; Cardiovascular; Hospitalizations; Death;
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GOLD B; OR GOLD E: Criteria: CAT ≥10 or MMRC ≥ 2 ; OR 2 exacerbations/year or 1 exacerbation leading to hospitalization
- GOLD 3 OR 4: Criteria: FVE1 < 50%

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is prevalent (8-20%) and is one of the leading causes of mortality. In 2019 according to WHO it was the third highest cause of death worldwide. In 2019 in Brazil respiratory diseases (Chapter J in the ICD10) were the third cause of death (176.073) with COPD (J44) accounting for 45.163 deaths (25,6% of respiratory and 3% overall). There is an upward trend for COPD mortality worldwide.

The disease also has a high morbidity leading to impairment in daily activity and quality of life.

Patients with severe and very severe disease are at a higher risk for negative outcomes, including exacerbation (up to 2-3 per patient per year). This in turn increases the risk of future exacerbations and mortality, with heightened risk lasting up to two years after each event. It is impertive to evaluate which sub-groups are at an even higher risk and could be potential targets for intervention.

"The PLATINO study" was conducted on 2004 and evaluated the prevalence of COPD in 5 cities, only one in Brazil - Sao Paulo. As the data is 20 years old it might not reflect the current epidemiological status and might not be representative of Brazil as a whole.

Understanding this population, their clinical and laboratorial characteristics can help identify sub-groups with higher risk and potential for intervention. The current prevalence, causing agent and characteristics are not known in Brazil as well as detailed outcome data.

DETAILED DESCRIPTION:
This is a prospective multicentre cohort, non-interventional study. The design is to have multiple medical centres representing the regions of Brazil. Each region has a different exposure to risk factors like tobacco smoke, biomass burning and environmental pollution, has a different population composition and density, degree of urbanization and education level. There are also some inferred genetic differences due to previous colonization and miscegenation. *CAT (COPD Assessment Test) OU CAAT (Chronic Airway Assesment Test).

The patients will be enrolled in non-random consecutive method and will be followed up for 12 months. There will be on-site visits at inclusion (V0), 6 and 12 months. There will tele-consults at 3 and 9 months to gather relevant clinical data, with special interest at exacerbation.

There will be 8 participating centres in Brazil, representing all 5 regions (North, Northeast, Midwest, Southeast and South). They will be Teaching Hospitals, Regional Reference Hospitals, Tertiary Hospitals or High Complexity Hospitals. The data will be collected on each site and will be adjudicated by the ARO Team.

ELIGIBILITY:
Inclusion Criteria:

Severe, very severe and symptomaitc COPD, according to GOLD definition: exposure, FEV1/FVC ratio <0,7:

* GOLD B (mMRC>=2, CAT>=10), OR
* GOLD E (>=2 moderate exacerbations or 1 severe), OR
* GOLD 3 and 4 (FEV1 <50%).

Exclusion Criteria:

Severe interstitial lung disease (extent >50% on HRCT), OR Severe pulmonary hypertension (on triple therapy), OR Active cancer - undergoing systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study will be adult patients, both sexes, with severe and very severe COPD enrolled in the participating centers.
Sampling Method: Probability Sample
Enrollment: 693 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of exacerbations, hospitalizations and death. | 12 months
  Rate of COPD exacerbations, hospitalizations and death.

SECONDARY OUTCOMES:
Clinical characteristics - GOLD grade (Global Intiative for Chronic Lung Disease) | 12 months
  Baseline and evolution of numeric and percentual data of the clinical characteristics: GOLD grade: Global Intiative for Chronic Lung Disease according to the 2024 guidelines (ABE, 1-4),
Clinical characteristics - spirometric parameters | 12 months
  Evolution of spirometric parameters (absolute in mL and % in relation to predicted). A higher value is better.
Clinical characteristics - BMI (Body mass index) | 12 months
  BMI: Body mass index (BMI - kg/m^2). Absolute number and division <=21 or >21.

OTHER OUTCOMES:
Incidence of exacerbations | 12 months
Incidence of non-fatal cerebrovascular and cardiovascular events | 12 months
Description of symptoms according to CAT score (COPD assessment test) | 12 months
  CAT: COPD assessment test score from 0-40, higher is more symptomatic.
Rate of decline in forced exprired volume in first second (FEV1) | 12 months
  Baseline to 12 months.
Description of quality of life score SGRQ-C (St. George Respiratory Questionaire - COPD) | 12 months
  SGRQ-C: St. George Respiratory Questionaire - COPD. The Total score is calculated by summing the weights to all the positive responses in each component. Score ranges from 0 to a Total (sum of maximum for all three components) 3201.9. Higher score is worse.
Description of symptoms according to mMRC (Modified Medical Research Council dyspnea scale) | 12 months
  mMRC: Modified Medical Research Council (dyspnea scale) 0-4, higher is worse
Description of symptoms 6MWT (6 minutes walk test) | 12 months
  6MWT: 6 minutes walk test (meters) 0-1000m, above 1000m is highly improbable, higher is better.
Description of treatment | 12 months
  Description of medication classes and dosages in use.
Clinical characteristics - laboratory data | 12 months
  Recent laboratory data will be analyzed and collected when available (e.g., eosinophils absolute count/mcL and %, IgE KU/L, chest CT report in pdf).

CONTACTS AND LOCATIONS:
Overall Officials: Henrique AR Fonseca, ScD, Study Chair — Hospital Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein (HIAE), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No